CLINICAL TRIAL: NCT00200928
Title: Asthma, a Disease Due to a Lack of Bacterial Infections in Childhood.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Asthma Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3.2.93.96.2
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-04-04 (Estimated); Status verified 2006-04

CONDITIONS: Food Allergy; Atopic Dermatitis; Asthma; Rhinitis
Keywords: prospective; randomised; intervention; BCG; atopy
MeSH Terms: conditions — Food Hypersensitivity; Dermatitis, Atopic; Asthma; Rhinitis

INTERVENTIONS:
Biological: BCG

SUMMARY:
The degree of TH1-skewing by mycobacteria is controlles by NRAMP1 gene polymorphisms and related to the degree of inhibition of TH2-mediated disease.

DETAILED DESCRIPTION:
A randomised single blinded intervention study in high-risk newborns vaccinated at the age of 6 weeks with BCG or placebo.

Inclusion: high-risk was defined as either a mother or a father and a sibling with present or past atopic disease.

Exclusion: maternal infection in the last week of pregnancy, the use of immunomodulatory drugs or antibiotics during pregnancy (mother), the use of antibiotics directly post-partum (newborn)

ELIGIBILITY:
Inclusion Criteria:

high-risk was defined as either a mother or a father plus a sibling with present or past atopic disease.

Exclusion Criteria:

maternal infection in the last week of pregnancy, the use of immunomodulatory drugs or antibiotics during pregnancy (mother) or directly post partum (newborn)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1999-01; Study Completion 2005-07

PRIMARY OUTCOMES:
Incidence and severity of atopic disease.

SECONDARY OUTCOMES:
SCORAD, lung function, IgE, cytokine production by PBMNC's, NRAMP-polymorphisms.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten O Hoekstra, MD PhD, Principal Investigator — Wilhelmina Children's Hospital Utrecht (UMCU)
Locations (1):
- Wilhelmina Children's Hospital (UMCU), Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: click for more information: Indiaan onderzoek — http://www.kinderallergologie.nl/